CLINICAL TRIAL: NCT00871676
Title: Use of Chewing Gum to Facilitate Appetite Control and Weight Loss in Overweight Individuals Treated by Lifestyle Modification
Brief Title: Use of Chewing Gum to Facilitate Appetite Control and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Kathleen McMahon, Ph.D, RD, William Wrigley Jr. Company
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 804361
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2009-03

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Behavior Therapy; Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Overweight/obese individuals being treated with lifestyle modification to facilitate weight loss.
  Interventions: Behavioral: Lifestyle modification
- 2 (Experimental): Lifestyle modification plus use of chewing gum to facilitate weight loss in overweight/obese persons.
  Interventions: Behavioral: Lifestyle modification plus gum

INTERVENTIONS:
Behavioral: Lifestyle modification — 16 weekly followed by 8 monthly group behavioral weight loss sessions.
  Other Names: Behavior modification; Behavioral weight loss
  Arms: 1
Behavioral: Lifestyle modification plus gum — 16 weekly followed by 8 monthly group behavioral weight loss sessions. Subjects were also given gum along with instructions for times and occasions to chew with the aim of facilitating weight loss and appetite control.
  Other Names: Behavior modification; Behavioral weight loss
  Arms: 2

SUMMARY:
This purpose of this study was to test the use of chewing gum as an adjunct to lifestyle modification to facilitate appetite control and weight loss in overweight and obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* 21-75 years of age
* Body Mass Index of 25-45 inclusive

Exclusion Criteria:

* major medical psychiatric conditions
* medications know to effect weight
* full or partial dentures
* 18 or fewer teeth
* regular gum chewing (≥ 2 pieces/day)
* use of any tobacco product
* sensitivity to the following ingredients (mint, magnolia bark, eggs, or English Muffins)
* history of PKU
* sensitivity or allergy to aspartame
* current/history of alcohol abuse or addiction (within 5 year)
* recreational drug use
* recent significant weight change (+/- 5% in previous 6 months)
* currently pregnant or nursing and willingness not to get pregnant during course of study
* participation in any other research studies
* proximity to clinic (within one hour)
* access to reliable transportation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | Week 16 and 52

SECONDARY OUTCOMES:
Appetite control | Weeks 4, 8, 12, 16 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wadden, Ph.D, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States